CLINICAL TRIAL: NCT02094040
Title: Effect of Municipality-based Post-discharge Follow-up Visit Including the Primary Physician on Early Re-hospitalization in High Risk People of 65+ Years. A Randomised Controlled Trial.
Brief Title: Municipality-based Post-discharge Follow-up Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holbaek Sygehus (Other)
Collaborators: Region Sjælland (Other); Danish Institute for Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3800H0.52-0059
Record Dates: First submitted 2014-03-12; First posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Frailty; Readmission; Transition; Primary Care
Keywords: frailty; readmission; transition; discharge; primary care
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follow-up visit (Experimental): Receive municipality-based follow-up visit including primary physician.
  Interventions: Behavioral: Receive municipality-based follow-up visit
- Usual care (No Intervention): Does not receive follow-up visit

INTERVENTIONS:
Behavioral: Receive municipality-based follow-up visit — Systematic electronic referral from hospital to municipality of high risk people at discharge from a medical ward. Contact from municipality service to primary physician and citizen, to arrange first home visit within 7 days with focus on: medication, rehabilitation plan and health care appointments, functional level and need for further health care initiatives. The visit is concluded by planning of further visits (up till tree) and division of responsibilities between primary physician and the municipality service.
  Other Names: Intervention group
  Arms: Follow-up visit

SUMMARY:
The purpose of this study is to determine whether discharge follow-up visit by primary physician and community-based nurse affects the risk of early re-hospitalisation among high risk older people discharged from a medical ward.

ELIGIBILITY:
Inclusion Criteria:

* Patient geography (The participant live in; Holbæk Kommune, Odsherred Kommune or Kalundborg Kommune.)
* Discharged from medical ward Holbæk Sygehus.
* Frailty (Rated by following criterion: dementia or a minimum of two of the following conditions; two or more hospitalisations within 12 month prior to follow up, los of physical function, treatment of two or more concurrent medical and/or surgical conditions, psychiatric disease, multi-pharmacy of more than 6 prescription medication, suspicious of congenital disturbances, substance abuse problem, disadvantaged social network, need for increasing home care following index hospitalization.)

Exclusion Criteria:

* Not discharged to home (If the patient are not discharged to home.)
* No written consent (If the patient does not wish to participate / written consent are not signed.)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 531 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Re-admission | Within 30 days from discharge
  The primary outcome is re-hospitalisation rate within 30 days from discharge. Data is obtained from the official register of danish patients (Landspatientregistret).

SECONDARY OUTCOMES:
Long-term hospitalization rate | Within 180 days from discharge
  Secondary outcome concerns hospitalization rate measured at 30 and 180 days post discharge. Data is obtained from the official register of Danish patients (Landspatientregistret).

OTHER OUTCOMES:
Long-term death rate | Within 180 days from discharge
  Other pre-specified outcome concerns death rate measured at 30 and 180 days post discharge. Data is obtained from the official register of Danish patients (Landspatientregistret).
Long-term use of primary health care services | Within 180 days from discharge
  Other pre-specified outcome concerns the use of primary health care services measured at 30 and 180 days post discharge. Data is obtained from the official register of primary health care in Denmark (Sygesikringsregistret) and registration from 3 Danish municipalities.
Long-term use of secondary health care services | Within 180 days from discharge
  Other pre-specified outcome concerns the use of secondary health care services measured at 30 and 180 days post discharge. Data is obtained from the official register of Danish patients (Landspatientregistret).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gjørup, Principal Investigator — Medicinsk Afdeling, Holbæk Sygehus
Locations (1):
- Medicinsk Afdeling, Holbæk Sygehus, Holbæk, Denmark

REFERENCES:
- [Derived] Thygesen LC, Fokdal S, Gjorup T, Taylor RS, Zwisler AD; Prevention of Early Readmission Research Group. Can municipality-based post-discharge follow-up visits including a general practitioner reduce early readmission among the fragile elderly (65+ years old)? A randomized controlled trial. Scand J Prim Health Care. 2015 Jun;33(2):65-73. doi: 10.3109/02813432.2015.1041831. Epub 2015 Jun 10. PMID 26059872